CLINICAL TRIAL: NCT00412906
Title: Study of Gene Expression in Fat and Muscle Tissue in Type 2 Diabetics and Healthy Controls During Experimental Endotoxemia
Brief Title: Study of Gene Activity in Fat and Muscle in Diabetics and Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Centre of Inflammation and Metabolism, Rigshospitalet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DM2.sa.cim.rh.dk
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Healthy; Type 2 Diabetes; Endotoxemia
Keywords: Low-grade inflammation; insulin resistance; Metabolism; Type 2 diabetes; Endotoxemia; Fat tissue; Muscle tissue; RT-PCR
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Endotoxemia; Insulin Resistance | interventions — endotoxin, Escherichia coli

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Escherichia Coli Endotoxin

SUMMARY:
The aim of the present protocol is to study gene activity in fat and muscle tissue in type 2 diabetics and healthy volunteers after injection of E. coli endotoxin.We hereby hope to gain insight in some mechanisms behind the association between inflammation and insulin resistance.

DETAILED DESCRIPTION:
Numerous studies have shown an association between low-grade inflammation and insulin-resistance in type 2 diabetics. It is also well-known that septic patients often develop insulin-resistance. The pathogenetic mechanisms behind the association between inflammation and insulin-resistance is not fully understood.

In this study we create an experimental inflammation by giving E. coli endotoxin 0,3 ng/kg iv to type 2 diabetics and healthy controls. Muscle biopsies are taken at 0, 2, 4 and 6 hours after injection, while fat biopsies are taken 0, 2, 4, 6 and 8 hours after endotoxin. mRNA for adiponectin, leptin, PPAR-gamma, PGC-1, PAI-1 and cytokines in tissue is later measured by RT-PCR.

Blood samples are drawn on an hourly basis until 8 hours after endotoxin injection for common biochemical analyses including white blood cell count. Plasma is spared and later analyzed for cytokines, PAI-1 and VCAM-1/ICAM-1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Type 2 diabetes

Exclusion Criteria:

* Heart failure
* Lung disease
* Anti-coagulation treatment

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Gene expression evaluated by measuring mRNA via RT-PCR. Plasma cytokine content, PLasma PAI-1 content, endotoxemia score

SECONDARY OUTCOMES:
Mean Arterial Pressure, heart rate, Temperature,

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sofie Andreasen, MD, Principal Investigator — Rogshospitalet, Denmark
Locations (1):
- Centre of Inflammaiton and Metabolism, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Andreasen AS, Kelly M, Berg RM, Moller K, Pedersen BK. Type 2 diabetes is associated with altered NF-kappaB DNA binding activity, JNK phosphorylation, and AMPK phosphorylation in skeletal muscle after LPS. PLoS One. 2011;6(9):e23999. doi: 10.1371/journal.pone.0023999. Epub 2011 Sep 13. PMID 21931634